CLINICAL TRIAL: NCT06812793
Title: Do Children With Cystic Fibrosis Differ in Muscle Endurance? A Comparative Study
Brief Title: Muscle Endurance in Children With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Betül Çınar, Lecturer, PhD, Bezmialem Vakif University
Other Study IDs: bvubcinar02
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
Keywords: Pediatric chest diseases; core muscle endurance; respiratory muscles; sit-to-stand test
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with cystic fibrosis: Children diagnosed cystic fibrosis
  Interventions: Other: Measurement of Core Muscle Endurance; Other: Respiratory Muscle Strength; Other: Respiratory Muscle Endurance; Other: Peripheral Muscle Endurance
- Healthy children: Age-matched healthy volunteers
  Interventions: Other: Measurement of Core Muscle Endurance; Other: Respiratory Muscle Strength; Other: Respiratory Muscle Endurance; Other: Peripheral Muscle Endurance

INTERVENTIONS:
Other: Measurement of Core Muscle Endurance — Endurance of the flexor, extensor and lateral trunk muscles will be assessed using the McGill Trunk Endurance Tests.
Other: Respiratory Muscle Strength — Inspiratory and expiratory muscle strength will be made with a portable, electronic intra-oral pressure measuring device.
Other: Respiratory Muscle Endurance — Respiratory muscle endurance testing will be measured using an inspiratory muscle training device at increasing threshold load.
Other: Peripheral Muscle Endurance — Peripheral muscle endurance will be assessed by performing 30 and 60 second sit-to-stand tests.

SUMMARY:
Cystic fibrosis (CF) is a genetic disorder affecting exocrine glands, leading to thick, viscous secretions that damage organs such as the lungs, pancreas, and reproductive system. Respiratory failure from CF lung disease is a major cause of morbidity and mortality, with chronic inflammation and infections disrupting mucociliary clearance. This results in declining respiratory functions, muscle strength, physical inactivity, and quality of life. While some studies compare respiratory and lower extremity muscle endurance in children with CF, none have evaluated core muscle endurance. This study aims to compare respiratory muscle strength, endurance, and muscle endurance in the core and lower extremities between children with CF and healthy peers.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an autosomal recessive genetic disease characterized by the involvement of exocrine glands, resulting from a disorder in the synthesis or function of the Cystic Fibrosis Transmembrane Regulator (CFTR) protein. The CFTR protein is responsible for ion and water transport in the cell epithelium. Dysfunction of this protein causes the secretion produced to be deficient in water. Viscous secretion, which is difficult to remove from its environment, causes permanent damage to many organs and systems such as the lungs, pancreas, hepatobiliary system and reproductive system. Respiratory failure due to CF lung disease is the most important cause of morbidity and mortality. The basic mechanism in the pathophysiology of CF lung disease is chronic inflammation and recurrent infections that occur as a result of the disruption of mucociliary clearance by sticky secretions. This vicious cycle causes obstruction in the airways and leads to progressive losses in respiratory functions. The decrease in respiratory functions; loss of muscle strength, reduced functional capacity, physical inactivity and reduced quality of life. There are limited studies in the literature comparing the respiratory muscle strength, respiratory muscle endurance and lower extremity muscle endurance of children with CF with their healthy peers. However, there is no study evaluating the core muscle endurance of children with CF. This study aims to compare the respiratory muscle strength, respiratory muscle endurance, core muscle endurance and lower extremity muscle endurance in children with CF and their healthy peers.

ELIGIBILITY:
Inclusion Criteria for Children with Cystic Fibrosis

* Being between the ages of 6-18,
* Being diagnosed with Cystic Fibrosis according to the American Cystic Fibrosis Association consensus guideline,
* Having a forced expiratory volume in one second (FEV1) above 40% of the predicted value

Exclusion Criteria for Children with Cystic Fibrosis

* Not being able to cooperate with the assessment methods performed in the study
* Having an orthopedic, neurological, vestibular, etc. problem that may negatively affect the assessment methods performed in the study
* Having a history of exacerbation in the last month
* Having an organ transplantation history
* Using systemic corticosteroids

Inclusion Criteria for Healthy Children

- Being between the ages of 6-18

Exclusion Criteria for Healthy Children

* Not being able to cooperate with the assessment methods performed in the study
* Having an orthopedic, neurological, vestibular, etc. problem that may negatively affect the assessment methods performed in the study
* Having had a respiratory tract infection in the last month

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children diagnosed with cystic fibrosis and age matched healthy volunteers who do not have any diagnosed chronic diseases
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Core muscles endurance | Baseline
  Endurance of the flexor, extensor and lateral trunk muscles will be assessed using the McGill Trunk Endurance Tests.

SECONDARY OUTCOMES:
Respiratory Muscle Strength | Baseline
  Inspiratory and expiratory muscle strength will be made with a portable, electronic intra-oral pressure measuring device.
Respiratory muscle endurance | Baseline
  Respiratory muscle endurance testing will be measured using an inspiratory muscle training device at increasing threshold load.
Peripheral muscle endurance | Baseline
  Peripheral muscle endurance will be assessed by performing 30 and 60 second sit-to-stand tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No